CLINICAL TRIAL: NCT01256775
Title: A Multicenter, Double-blind, Randomized, Parallel Group Study to Assess the Effect of NCX4016 vs Placebo on Walking Distance in Patients With Peripheral Arterial Occlusive Disease at Leriche-Fontaine Stage II
Brief Title: Effect of NCX4016 on Walking Distance in Patients With Peripheral Arterial Occlusive Disease (PAOD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NicOx Research Institute S.r.l. (Industry)
Responsible Party: NicOx Research Institute, Paolo Gresele, University of Perugia - Italy
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NCX4016-X-208
Record Dates: First submitted 2010-12-06; First posted 2010-12-09 (Estimated); Last update posted 2011-01-19 (Estimated); Status verified 2011-01

CONDITIONS: Intermittent Claudication
Keywords: atherosclerosis; carotid intima-media thickness; intermittent claudication; Nitric Oxide / NO
MeSH Terms: conditions — Intermittent Claudication; Atherosclerosis | interventions — nitroaspirin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NCX4016 placebo (Placebo Comparator): NCX4016 placebo b.i.d for 6 months
  Interventions: Drug: NCX4016 placebo
- NCX4016 (Active Comparator): ncx4016,800 mg b.i.d., on top of aspirin 100 mg o.d.
  Interventions: Drug: NCX-4016

INTERVENTIONS:
Drug: NCX-4016 — NCX4016 800 mg b.i.d. for 6 months on top of aspirin 100 mg o.d.
  Arms: NCX4016
Drug: NCX4016 placebo — NCX4016 placebo b.i.d. for 6 months
  Arms: NCX4016 placebo

SUMMARY:
Peripheral arterial disease (PAD) is almost invariably associated with a generalized atherosclerotic involvement of the arterial tree and endothelial dysfunction. Previous short term studies showed improvement of vascular reactivity and walking capacity in PAD patients by measures aimed at restoring Nitric Oxide (NO) production. NO is also known to prevent the progression of atherosclerosis. We wished to assess whether the prolonged administration of a NO-donating agent (NCX 4016) improves the functional capacity of PAD patients and affects the progression of atherosclerosis as assessed by carotid intima-media thickness (IMT).

Four hundred forty two patients with stable intermittent claudication were enrolled in a prospective, double blind, placebo-controlled study and randomized to either NCX 4016 800mg bid or its placebo for 6 months. The primary study outcome was the absolute claudication distance (ACD) on a constant treadmill test (10% incline, 3km/hr); main secondary end-point was the change of the mean far-wall right common carotid artery IMT.

DETAILED DESCRIPTION:
Design of the study This was a prospective, randomized, double-blind, parallel-groups, placebo-controlled study conducted in fortythree clinical sites throughout Europe. 442 patients with peripheral arterial occlusive disease (PAD) at Leriche-Fontaine stage II were treated with NCX 4016 800 mg bid or with an indistinguishable placebo for 6 months. The dosage of 800 mg bid was selected based on previous clinical studies, which demonstrated a good safety profile and a good tolerability in the gastro intestinal tract. Compliance was checked by counting dispensed versus returned study medication.

All patients received 100 mg aspirin once daily for cardiovascular prevention, standard for this patient population at the time of study design.

Inclusion criteria were: male and female patients between 40 and 80 years with Leriche-Fontaine stage II PAD presenting symptoms of intermittent claudication stable for at least 6 months, an ankle/brachial index <0.9, an absolute claudication distance (ACD) <500 m and an initial claudication distance (ICD) >50 m on a standardized treadmill test (3% incline, 3 km/hr), and clinical stability before inclusion (i.e. changes in ACD not exceeding 25% in two standardized treadmill tests during run-in). All patients gave their written informed consent.

Exclusion criteria were: unstable symptoms and/or rapid deterioration of PAD during the previous 3 months; presence of clinically significant renal or hepatic failure, or insulin-dependent type 1 diabetes; uncontrolled type 2 diabetes, arterial hypertension or dyslipidemia; any clinical condition limiting the patient's exercise ability (angina pectoris, congestive heart failure, respiratory disease, bone and joint disease, neurological disorders); active peptic ulcer during the previous 6 months; any hemorrhagic condition or history of bleeding; acute coronary syndrome or acute cerebrovascular episodes during the previous 6 months; previous revascularization procedures during the last 6 months or indication for vascular surgery; ischemic rest pain; life expectancy <12 months; pregnancy or lactation; participation to other investigational trials within 3 months prior to inclusion; history of hypersensitivity or any form of allergic reaction or contraindications to NSAIDs, aspirin, and NO-donating drugs. The following treatments were not allowed for the period of the study: continuative use (>7 days) of NSAIDs or nitrovasodilating drugs; phosphodiesterase type 5 inhibitors, anticoagulants, heparin, ticlopidine, clopidogrel, indobufen, defibrotide, mesoglycan, picotamide, pentoxyfylline, carnitine, sulodexide. All other concomitant treatments were kept constant as much as possible during the study period.

Primary end-point of the study was the ACD on a constant treadmill test; secondary end-points were ICD; responder rates, i.e. the proportion of patients showing a >=28% or a >=50% improvement of ACD in comparison with baseline; quality of life questionnaire Short-Form 36 (SF-36); the variations of the ankle/brachial index (ABI) between baseline and 6 months and the modifications of the intimal medial thickness (IMT) of the common right carotid artery at 6 months as compared with baseline.

Common right carotid artery was examined by B-mode ultrasound in the longitudinal view, 1-1.5 cm proximally to the bifurcation. The measurement of IMT was obtained according to the Mannheim carotid intima-media thickness consensus with one modification: instead of acquiring the vascular wall image only with the lateral probe incidence, images were acquired also with the anterior and posterior incidence, in order to obtain a triplicate number of measurements to be used for comparisons. Each position was visualized and recorded for at least 15 sec. with simultaneous taking of the ECG tracing. Images of the far wall of the distal 1 cm of the right common carotid artery were obtained. IMT was calculated from each of the three projections and the final value was calculated from the average of all measurements with the use of standardized ultrasonography settings. The baseline carotid ultrasonographic examinations were used to localize the site of interest at follow-up. Digitized still images from an electrocardiographically defined diastolic frame were analyzed offline. A single observer who was unaware of the treatment assignments and the identities of the patients measured the mean carotid intima media thickness. Focal atherosclerotic plaques were excluded from the measurements. All measurements were performed with the use of an automated border detection system. A number of measurements not inferior to 30 for each of the three image acquisition incidences was carried out in the 1cm segment of the carotid artery assessed. For each subject the same ultrasound system and transducer and the same operator were used throughout the study. Images were centrally analyzed at the coordinating center by a dedicated, automated computerized edge detection system for the measurement of common carotid far wall intima-media using the software M'ATH 2.0 (Metris Argenteuil, France).

ELIGIBILITY:
Inclusion Criteria:

* male and female patients between 40 and 80 years with Leriche-Fontaine stage II PAD presenting symptoms of intermittent claudication stable for at least 6 months
* ankle/brachial index <0.9
* an absolute claudication distance (ACD) <500 m
* an initial claudication distance (ICD) >50 m on a standardized treadmill test (3% incline, 3 km/hr)
* and clinical stability before inclusion (i.e. changes in ACD not exceeding 25% in two standardized treadmill tests during run-in).
* all patients gave their written informed consent.

Exclusion Criteria:

* unstable symptoms and/or rapid deterioration of PAD during the previous 3 months
* presence of clinically significant renal or hepatic failure, or insulin-dependent type 1 diabetes
* uncontrolled type 2 diabetes, arterial hypertension or dyslipidemia
* any clinical condition limiting the patient's exercise ability (angina pectoris, congestive heart failure, respiratory disease, bone and joint disease, neurological disorders)
* active peptic ulcer during the previous 6 months
* any hemorrhagic condition or history of bleeding
* acute coronary syndrome or acute cerebrovascular episodes during the previous 6 months
* previous revascularization procedures during the last 6 months or indication for vascular surgery; ischemic rest pain
* life expectancy <12 months
* pregnancy or lactation
* participation to other investigational trials within 3 months prior to inclusion
* history of hypersensitivity or any form of allergic reaction or contraindications to NSAIDs, aspirin, and NO-donating drugs
* the following treatments were not allowed for the period of the study: continuative use (>7 days) of NSAIDs or nitrovasodilating drugs
* phosphodiesterase type 5 inhibitors, anticoagulants, heparin, ticlopidine, clopidogrel, indobufen, defibrotide, mesoglycan, picotamide, pentoxyfylline, carnitine, sulodexide
* All other concomitant treatments were kept constant as much as possible during the study period.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 442 (Actual)
Dates: Start 2003-09; Primary Completion 2005-04 (Actual); Study Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
maximal walking distance evaluated by a constant treadmill test | baseline
maximal walking distance evaluated by a constant treadmill test | 6 months

SECONDARY OUTCOMES:
pain-free walking distance | baseline, 1-3-6 months
assessment of carotid artery IMT | baseline and 6 month

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Gresele, M.D., Ph.D., Principal Investigator — University Of Perugia
Locations (1):
- Ospedale di Perugia, Perugia, Italy, Italy